CLINICAL TRIAL: NCT06457802
Title: A Multiple Technology-Based and Individually Tailored Sit Less Program for Patients With Type 2 Diabetes: A Randomized Controlled Trial
Brief Title: Sit Less Program for Patients With Type 2 Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI terminated the study due to unforeseen extenuating personal circumstances. The VUMC IRB approved the early termination of the study on 8/20/2024. The last day the participants received the intervention was 08/20/2024.
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Shelagh Mulvaney, Principal Investigator, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 240549
Record Dates: First submitted 2024-05-28; First posted 2024-06-13 (Actual); Results first posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes; Sedentary Behavior; Sedentary Time; Physical Activity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study employs a parallel assignment interventional model, wherein participants are randomly allocated to one of two groups: the intervention group or the control group. The intervention group will receive a comprehensive sedentary behavior (SB) reduction program over 8 weeks, utilizing wearable technology, including Fitbit devices and smart water bottles, combined with personalized text message prompts. The control group will receive standard care, consisting of educational materials provided by the American Heart Association, without additional prompts or interventions. The primary goal is to compare the outcomes between these two groups to assess the feasibility, acceptability, and preliminary efficacy of the SB reduction intervention in reducing SB and improving cardiometabolic health and patient-centered outcomes in individuals with type 2 diabetes.
Who Masked: Outcomes Assessor
Masking Description: Single-blind; The participants and the interventionists will be aware of the treatment assignments, but the data collectors will be blinded to the group assignments to reduce bias in data collection and analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sit Less Group - mHealth intervention (Experimental): The intervention group will target a 120 minute per day reduction in sedentary behavior using an objective activity monitor and mHealth. Outcomes will be measured at baseline and post-intervention.
  Interventions: Behavioral: Sit Less Program
- Control Group - Standard Care (No Intervention): Participants in the control group will receive standard care, including educational materials from the American Heart Association's Healthy Living booklet and a Fitbit. They will not receive the smart water bottle or the tailored text messages aimed at reducing sedentary behavior. The Fitbit move alert setting will be disabled for the control group.

INTERVENTIONS:
Behavioral: Sit Less Program — The intervention group will target a 120 minute per day reduction in sedentary behavior using an objective activity monitor and mHealth. Outcomes will be measured at baseline and post-intervention.
  Arms: Sit Less Group - mHealth intervention

SUMMARY:
This randomized controlled trial aims to evaluate an 8-week intervention designed to reduce sedentary behavior (SB) in patients with type 2 diabetes (T2D) using wearable technology. The intervention involves the use of Fitbit devices to prompt standing/walking breaks, a smart water bottle to encourage hydration-related movement, and tailored text messages for behavior reinforcement. Participants will be assessed at baseline and post-intervention for changes in SB, light physical activity, cardiometabolic markers, and patient-centered outcomes. The study seeks to determine the intervention's acceptability and preliminary efficacy in reducing SB and improving health outcomes in T2D patients.

DETAILED DESCRIPTION:
The investigators propose to develop and conduct a pilot randomized controlled trial to test a wearable technology-based sedentary behavior (SB) reduction intervention in type 2 diabetes (T2D) patients. The study will recruit 80 participants who will be randomized to either the control group or the intervention group. The 8-week intervention aims to reduce daily SB by at least 120 minutes through the use of Fitbit devices, a smart water bottle, and tailored text messages. Participants will set personalized SB reduction goals and receive prompts to stand or walk, along with hydration reminders from the smart water bottle to encourage movement.

Specifically, the study aims to: determine the acceptability of the SB reduction intervention in T2D patients by evaluating satisfaction and compliance; evaluate the preliminary efficacy of the intervention on reducing total SB time and numbers of prolonged SB bouts; and explore preliminary effects on light physical activity, cardiometabolic markers (24-hour glycemic control, BMI, waist circumference, blood pressure), and patient-centered outcomes (confidence in reducing SB, habit strength for SB, and quality of life). Outcomes will be measured at baseline and post-intervention using biometric assessments, questionnaires, and continuous glucose monitoring. The study seeks to provide insights into the feasibility and potential health benefits of a technology-driven SB reduction program for T2D patients.

ELIGIBILITY:
Inclusion Criteria:

* ages 18 and above
* diagnosed with type 2 diabetes
* self-reported HbA1C<13
* self-report of sitting ≥ 8hr/day
* ability to stand and walk
* ownership of a smartphone.

Exclusion Criteria:

* currently using an activity tracker
* currently participating in exercise or other research programs.
* random blood glucose > 300 mg/dL.
* non-English speaking.
* patients classified as unstable (e.g., heart failure, uncontrolled arrhythmia) or have kidney disease that limits daily water intake.
* any conditions that prevent standing or walking due to physical or cognitive limitations, such as cognitive impairment, severe pain, problems with lower limbs, or a history of surgeries that limit movement.
* participation in Sit Less Program V1 (IRB #221566).
* currently pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2024-06-12 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shelagh Mulvaney, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sit Less Group - mHealth Intervention | Control Group - Standard Care
Started | 2 | 2
Completed | 0 | 0
Not Completed | 2 | 2
Not completed — Early termination of study prior to participant completion | 2 | 2

BASELINE CHARACTERISTICS:
Population: No data analyzed. As only 4 participant were enrolled in this study, no data is reported here, in order to protect and maintain participant privacy/confidentiality.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sit Less Group - mHealth Intervention | Control Group - Standard Care | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Customized [Mean (Full Range); unit: years]
  Age (Mean and Range) | 62.0 [58 to 68] | 57.5 [42 to 73] | 59.75 [42 to 73]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/Gender (Count): Female | 2 | 2 | 4
  Sex/Gender (Count): Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity (Count): White (Not Hispanic or Latino) | 2 | 1 | 3
  Race/Ethnicity (Count): Hispanic or Latino | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4
Baseline Total Sedentary Behavior Time [Mean (Standard Deviation); unit: minutes/day] — Sedentary behavior will be objectively measured using the activPAL device, which participants will wear on their thigh for 7 days at both baseline and post-intervention. The activPAL device will record the amount of time (minutes/day) participants spend sitting or lying down during waking hours each day.
  minutes/day | 616.39 (61.96) | 616.39 (61.96) | 616.39 (61.96)

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Sedentary Behavior Time
Description: The primary outcome measure will assess the change in total sedentary behavior (SB) time from baseline to post-intervention. Sedentary behavior will be objectively measured using the activPAL device, which participants will wear on their thigh for 7 days at both baseline and post-intervention. The activPAL device will record the amount of time participants spend sitting or lying down during waking hours each day.
Time Frame: Baseline and 8 weeks post-intervention
Population: Zero participants completed the study. Change was not assessed as no data was collected for this outcome measure at 8-weeks post intervention.
Arm/Group | Sit Less Group - mHealth Intervention | Control Group - Standard Care
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Acceptability of the Sedentary Behavior Reduction Intervention
Description: Satisfaction will be assessed using a 23-item questionnaire. This questionnaire includes items on the perceived helpfulness, ease of use, and overall experience with the wearable devices, text messages, and goal-setting sessions. The questionnaire uses a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate greater satisfaction with the intervention.
Time Frame: 8 weeks post-intervention
Population: Zero participants completed the study. Data was not collected for this outcome measure as no questionnaires were completed 8-weeks post intervention.
Arm/Group | Sit Less Group - mHealth Intervention | Control Group - Standard Care
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Usability of the Sedentary Behavior Reduction Intervention
Description: Usability will be assessed using a 10-item System Usability Scale. The System Usability Scale provides a global measure of usability and uses a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). It has a minimum score of 0 and a maximum score of 100, where higher scores indicate better usability.
Time Frame: 8 weeks post-intervention
Population: as for outcome 2
Arm/Group | Sit Less Group - mHealth Intervention | Control Group - Standard Care
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Compliance With the Sedentary Behavior Reduction Intervention - Fitbit Usage
Description: Compliance with the intervention will be evaluated by tracking the usage data from the Fitbit devices, specifically the number of days the device was worn for at least 10 hours per day.
Time Frame: 8 weeks post-intervention
Population: as for outcome 2
Arm/Group | Sit Less Group - mHealth Intervention | Control Group - Standard Care
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Adherence to Sedentary Behavior Goals
Description: Adherence will be evaluated by tracking the percentage of set sedentary behavior reduction goals met by participants.
Time Frame: 8 weeks post-intervention
Population: as for outcome 2
Arm/Group | Sit Less Group - mHealth Intervention | Control Group - Standard Care
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Response Rates to Tailored Text Messages
Description: Compliance will be evaluated by tracking the response rates (percentage) to the tailored text messages sent as part of the intervention.
Time Frame: 8 weeks post-intervention
Population: as for outcome 2
Arm/Group | Sit Less Group - mHealth Intervention | Control Group - Standard Care
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Number of Prolonged Sedentary Bouts
Description: This measure will assess the change in the number of prolonged sedentary bouts, defined as periods of uninterrupted sitting or lying down lasting 30 minutes or more. Data will be collected using the activPAL device worn by participants for 7 days at both baseline and post-intervention.
Time Frame: Baseline and 8 weeks post-intervention
Population: as for outcome 1
Arm/Group | Sit Less Group - mHealth Intervention | Control Group - Standard Care
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Light Physical Activity
Description: This measure will evaluate changes in light physical activity, including total standing and stepping times. Participants will wear the activPAL device for 7 days at both baseline and post-intervention to capture these activity levels.
Time Frame: Baseline and 8 weeks post-intervention
Population: as for outcome 1
Arm/Group | Sit Less Group - mHealth Intervention | Control Group - Standard Care
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in 24-Hour Glycemic Control (GMI)
Description: 24-hour glucose levels will be measured by continuous glucose monitoring over a 7-day period. The 24-hour glucose control will be evaluated using the Glucose Management Indicator (GMI), which provides an estimated average glucose (eAG) based on the mean 24-hour glucose levels. The GMI will be calculated from the mean glucose values and reported as a single aggregated value. Additionally, the numbers of events and time in hypoglycemia (glucose < 3.9 mmol/L), euglycemia (glucose 3.9-7.8 mmol/L), hyperglycemia (glucose > 7.8 mmol/L), and above target (glucose > 9 mmol/L) will be monitored to provide context to the GMI value, but these will not be separately reported as primary outcome measures.
  Unit of Measure: GMI (Glucose Management Indicator, as a percentage)
Time Frame: Baseline and 8 weeks post-intervention
Population: as for outcome 1
Arm/Group | Sit Less Group - mHealth Intervention | Control Group - Standard Care
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change in Body Mass Index (BMI)
Description: This measure will evaluate changes in BMI, calculated using participants' height and weight measurements taken at baseline and post-intervention.
Time Frame: Baseline and 8 weeks post-intervention
Population: as for outcome 1
Arm/Group | Sit Less Group - mHealth Intervention | Control Group - Standard Care
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change in Waist Circumference
Description: This measure will assess changes in waist circumference, measured at the narrowest point between the rib cage and the iliac crest using a flexible tape measure.
Time Frame: Baseline and 8 weeks post-intervention
Population: as for outcome 1
Arm/Group | Sit Less Group - mHealth Intervention | Control Group - Standard Care
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change in Blood Pressure
Description: This measure will evaluate changes in systolic and diastolic blood pressure, measured using an automated and validated blood pressure monitor at baseline and post-intervention.
Time Frame: Baseline and 8 weeks post-intervention
Population: as for outcome 1
Arm/Group | Sit Less Group - mHealth Intervention | Control Group - Standard Care
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change in Confidence in Reducing Sedentary Behavior
Description: This measure will assess changes in participants' confidence in their ability to reduce sedentary behavior, evaluated using a validated self-efficacy questionnaire for physical activity and sedentary behavior. Confidence in reducing SB and increasing physical activity will be measured using 12 items from the Self-Efficacy Questionnaire for Physical Activity and Sedentary Behavior (Cronbach's alpha = 0.79). Each item is rated on a 5-point Likert scale ranging from 1 (not at all confident) to 5 (extremely confident). The total score ranges from 12 to 60, with higher scores indicating greater confidence in reducing sedentary behavior and increasing physical activity.
Time Frame: Baseline and 8 weeks post-intervention
Population: as for outcome 1
Arm/Group | Sit Less Group - mHealth Intervention | Control Group - Standard Care
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Change in Habit Strength for Sedentary Behavior
Description: This measure will evaluate changes in habit strength for sedentary behavior, assessed using the Self-Report Habit Index adapted for sedentary breaks (standing/walking). Habit strength for SB will be assessed by using a validated measure, Self-Report Habit Index (Cronbach's alpha = 0.91). This 7- item index was adapted to sedentary breaks (standing/walking) to assess the degree to which sedentary breaks become habitual. Each item is rated on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). The total score ranges from 7 to 35, with higher scores indicating stronger habit strength for taking sedentary breaks.
Time Frame: Baseline and 8 weeks post-intervention
Population: as for outcome 1
Arm/Group | Sit Less Group - mHealth Intervention | Control Group - Standard Care
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Change in Quality of Life
Description: Quality of life will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS)-Global Health, a 10-item measure developed by the NIH as an indicator for Healthy People. Each item is rated on a 5-point Likert scale, and the total score is calculated to range from 10 to 50. Higher scores indicate better quality of life.
Time Frame: Baseline and 8 weeks post-intervention
Population: as for outcome 1
Arm/Group | Sit Less Group - mHealth Intervention | Control Group - Standard Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Start of intervention for up to 8 weeks
Description: The definition of adverse event used in this study is consistent with the clinicaltrials.gov definition - any untoward medical occurrence associated with the use of an intervention, whether or not considered related to the intervention. Serious adverse events, as defined by the FDA, were not observed in this study.
Arm/Group | Sit Less Group - mHealth Intervention | Control Group - Standard Care
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-15): https://cdn.clinicaltrials.gov/large-docs/02/NCT06457802/Prot_SAP_000.pdf
  • Informed Consent Form (2024-06-03): https://cdn.clinicaltrials.gov/large-docs/02/NCT06457802/ICF_001.pdf